CLINICAL TRIAL: NCT05421000
Title: Assessing the Applicability and Potential Benefits of Wide Awake Local Anaesthesia No Tourniquet in Distal Radius Fracture Osteosynthesis.
Brief Title: WALANT in Distal Radius Fracture Osteosynthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Arnau de Vilanova (Other)
Collaborators: Institut de Recerca Biomèdica de Lleida (Other)
Responsible Party: Principal Investigator, Ana Scott-Tennent, Principal investigator. Orthopaedic surgeon in Upper Extremity department, Hospital Arnau de Vilanova
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CEIC-2360
Record Dates: First submitted 2022-06-01; First posted 2022-06-16 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Radius Fracture Distal
Keywords: Radius Fracture Distal; Local Anesthesia; Brachial Plexus Anesthesia; Osteosynthesis, Fracture
MeSH Terms: conditions — Wrist Fractures; Fractures, Bone | interventions — Tourniquets

STUDY DESIGN:
Intervention Model Description: Patients who had a surgical distal radius fracture, met all the inclusion criteria and signed the informed consent were randomized either to Group A in which WALANT technique was performed or Group B in which locoregional anesthesia(LRA) and upper limb tourniquet was used. This process was done by the external observer with 10 block randomization. Blinding was not possible as the differences between the anesthetic techniques are evident. However, none of the patients nor the surgeon or the anesthesiologist knew the group of intervention until the patient arrived at the operating anteroom the same day of surgery.
  Since the investigators considered this was a complex intervention, all patients were offered to receive sedation from the anesthesiologist if they presented any level of anxiety.
Who Masked: Participant, Care Provider
Masking Description: 10 block randomization was done by an external observer. Accordingly, the surgeon, the anesthesic or the patient didn't know about intervention until it was time to be exposed to the treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WALANT (Experimental): Wide awake local anesthesia without tourniquet was used for surgery
  Interventions: Procedure: WALANT
- Locoregional anesthesia and tourniquet (Active Comparator): Locoregional anesthesia (normally axillary block) and tourniquet was used for surgery
  Interventions: Procedure: Locoregional anesthesia and tourniquet

INTERVENTIONS:
Procedure: WALANT — Wide awake local anesthesia without tourniquet for distal radius fracture surgery
  Arms: WALANT
Procedure: Locoregional anesthesia and tourniquet — Locoregional anesthesia and tourniquet for distal radius fracture surgery
  Arms: Locoregional anesthesia and tourniquet

SUMMARY:
The purpose of this study is to assess the applicability and potential benefits of Wide Awake Local Anesthesia No Tourniquet (WALANT) or Local Anesthesia No Tourniquet ("LANT) versus locoregional anesthesia (LRA) and tourniquet in osteosynthesis of distal radius fractures (DRF) during the immediate postoperative period. Our hypothesis is that being able to avoid the use of a limb tourniquet in such a procedure may cause less swelling and better surgical wound appearance in the immediate postoperative period, without compromising pain level, patient satisfaction, or improving the number of complications. In this regard, prospective randomized study was designed comparing short term results of patients who were operated using WALANT (A) to locoregional anesthesia (LRA) and tourniquet (B). Main outcomes were pain, swelling and patient satisfaction. Surgical wound bleeding,mobility, surgeon's technical difficulty, insufficient anesthesia and complications were also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients who attended our hospital from December 2020th to December 2021 with DRF requiring surgical treatment who provided written informed consent and did not have any of the following excluding conditions described below

Exclusion Criteria:

1. Unsigned informed consent
2. 17 years old or younger
3. Associated fractures in which additional osteosynthesis was required: scaphoid fracture, ulnar fracture (ulnar styloid osteosynthesis included), bifocal radius fractures, etc
4. Open fractures
5. Polytrauma patients
6. Requiring more than a standard volar DRF approach and/or other than a volar plate.
7. DRF with >30 days or DRF malunions Contraindications to the use of ischemia

a. Peripheral vascular disease b. Extensive soft tissue injury c. Peripheral neuropathy d. Severe infection e. Thromboembolic disease in the extremity f. Poor skin conditions g. Arteriovenous fistula h. Sickle cell hemoglobinopathy

Contraindications for proximal blocking:

1. Existence of previous trauma or anatomical distortion of the area that prevents the abduction of the arm
2. Active presence of infection at the locoregional anesthesia puncture site
3. Previous axillary lymphadenopathy
4. Previous history of local anesthetic allergy
5. Severe coagulopathy
6. Severe pre-existing neurological diseases in the upper extremity

   Contraindications for WALANT anesthetic technique
7. Documented hypersensitivity to lidocaine
8. Compromised peripheral circulation
9. Patients with previous vascular pathology, a history of vasculitis, Buerger's disease, and scleroderma
10. Patients with infection of the area surrounding the injection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-12-20 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change between baseline patient's pain, immediately after the intervention, 24 hours after surgery, between 10 or 15 days after surgery and at 1 month after surgery | Baseline, 24 hours after surgery, between 10 and 15 days after surgery, 1 month follow up
  Pain using Visual Analogue Scale (VAS) scale and analgesia used (1 to 10 score. 10 means worst pain possible, 1 is almost no pain)
Change in baseline wrist swelling with 24 hours after surgery, between 10 or 15 days after surgery and at 1 month after surgery. | Baseline, 24 hours after surgery, between 10 and 15 days after surgery, 1 month follow up
  Difference between preoperative and postoperative swelling. Swelling was measured as Proximal wrist crease perimeter (cm). Healthy wrist was also measured to allow comparison.
Patient satisfaction | Written down in a questionnaire form delivered and answered by the patient between 10 and 15 days after surgery.
  Index of satisfaction, willingness to repeat and recommend the anesthetic technique. Personal designed "Satisfaction" scale (1 no satisfied- 5 very satisfied); 2 questions about whether he/she would repeat and recommend the anesthesia received (Yes/No answer)

SECONDARY OUTCOMES:
Evolution of active bleeding through surgical wound after surgery | 24 hours after surgery, between 10 and 15 days after surgery, 1 month follow up
  Presence of active bleeding through the surgical wound
Evolution in postoperative thumb mobility | 24 hours after surgery, between 10 and 15 days after surgery, 1 month follow up
  Kapandji scale for thumb mobility (1 to 10 scale. 10 represents the best thumb mobility and opposition possible, while 1 is almost no mobility)
Difficulty in visualization of surgical field | During surgery
  Asked by the external observer to the surgeon right after the surgery had finished. Personal scale (1 easy- 5 very difficult)
Stress during surgery | During surgery
  asked by the external observer to the surgeon right after the surgery had finished. Yes/no question and description of the reason of stress if any.
Number of complications after surgery | Collected at end of follow up (1 month)
  Description of complications regarding surgery or anesthetical technique
Evolution in postoperative finger mobility | 24 hours after surgery, between 10 and 15 days after surgery, 1 month follow up
  Capability to reach the distal and the proximal palmar crease with the tip of the fingers, named after 1st line and 2nd line respectively (according to intrinsic and extrinsic movement). If not arrived, the investigator's used the number of the observer's finger widths left to arrive each crease (i.e. 1 finger widths, 2 fingers widths)
Evolution of surgical wound bleeding after surgery | 24 hours after surgery, between 10 and 15 days after surgery, 1 month follow up
  Amount of blood encountered in the dressings (measured as on third, two thirds or more than two thirds of blood within the whole dressing/gauge)
Evolution in postoperative wrist mobility | 24 hours after surgery, between 10 and 15 days after surgery, 1 month follow up
  Flexion, extension, radial and ulnar deviation, pronation and supination using a goniometer (º)
Number of patients who need reconversion to general anaesthesia due to lack of effectiveness of anaesthetic technique | During surgery
  Yes or no answer to the question "does the patient need reconversion to general anaesthesia?"
Number of patients who need adding some extra anaesthesia due to lack of effectiveness of anaesthetic technique | During surgery
  Yes or no answer to the question "does the patient need extra anaesthesia?"
Description of reason why the patient needs adding some extra anaesthesia if necessary due to lack of effectiveness of the main anaesthetic technique | During surgery
  Open answer question describing the reason of anaesthesia insufficiency (for instance: pain, anxiety, discomfort, etc)
Type of anaesthetic technique added to solve the lack of effectiveness of the main anaesthesia | During surgery
  Open answer question describing the technique used in order to resolve lack of anaesthesia if needed (sedation, extra doses of local anaesthetic, anatomic location of local anaesthetic, doses of local anaesthetic, etc)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Scott-Tennent, Miss, Principal Investigator — Hospital Arnau Vilanova
Locations (1):
- Hospital Arnau Vilanova, Lleida, Segria, Spain

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-10): https://cdn.clinicaltrials.gov/large-docs/00/NCT05421000/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-10): https://cdn.clinicaltrials.gov/large-docs/00/NCT05421000/ICF_001.pdf